## Statistical Analysis Plan

## 1 Title page

Full Title Objective Randomised Blinded Investigation of Therapeutic

Ablation versus cardioversion for persistent Atrial

**Fibrillation** 

Short Title/Acronym ORBITA-AF Pilot Trial

Sponsor Queen Mary, University of London

Contact person of the above sponsor organisations is:

Dr Mays Jawad

**R&D** Operations Manager

Barts Health - QMUL Joint Research Management Office

(JRMO)

Queen Mary University of London 5 Walden Street, Whitechapel

London, E1 2EF

Phone: 020 7882 7275

Email: <a href="mailto:research.governance@qmul.ac.uk">research.governance@qmul.ac.uk</a>

REC Reference 19/LO/0775

IRAS Reference 237038

**ReDA Number** Not applicable

**Chief Investigator** Professor Richard Schilling

Principal Investigator Dr Malcolm Finlay

**Co-Investigator** Dr Vivienne Monk

**Designated Sites**Barts Heart Centre

# 2 SAP revision history

| Protocol Version | Updated SAP version No. | Section number changed | Description of and reason for change | Date changed |
|---|---|---|---|---|
| 5.0 | 1.0 | NA | NA | NA |
| 8.0 | 2.0 | 11.1 | Amendment to include an interim analysis, in line with the trial protocol. | 10 June 2022 |

# 3 Table of contents

| 1 | 7 | Γitle | e pa | ge | 1 |
|---|---|---|---|---|---|
| 2 | 5 | SAP | Sig | natures | |
| 3 | S | SAP | rev | ision history | 2 |
| 4 | ٦ | Гаb | le o | f contents | 3 |
| 5 | ( | GLC | SSA | ARY of Terms and Abbreviations | 5 |
| 6 | I | ntr | odu | ction | 6 |
| | 6.1 | | Pref | face | 6 |
| | 6.2 | 2 | Pur | pose of the analyses | 6 |
| 7 | 5 | Stuc | ly o | bjectives and design | 6 |
| | 7.1 | | Des | sign | 6 |
| | 7.2 | 2 | Stu | dy objectives | 6 |
| | 7.3 | 3 | Fea | sibility Endpoints | 7 |
| | 7.4 | 1 | Effi | cacy Endpoints | 7 |
| | 7 | 7.4. | 1 | Primary endpoint | 7 |
| | 7 | 7.4. | 2 | Secondary endpoints | 7 |
| | 7 | 7.4. | 3 | Schedule of Assessment | 8 |
| | 7 | 7.4. | 4 | Assessment of feasibility endpoints | 9 |
| | 7 | 7.4. | 5 | Assessment of primary and secondary effic | acy endpoints9 |
| | 7.5 | 5 | Lev | el of significance | 10 |
| | 7.6 | <b>;</b> | San | nple size | 10 |
| 8 | ( | Gen | eral | Analysis Definitions | 10 |
| | 8.1 | | Stu | dy period and visit definitions | 10 |
| | 8 | 3.1. | 1 | Visits | 10 |
| | 8 | 3.1. | 2 | Study Scheme Diagram | 12 |
| | 8.2 | 2 | Stu | dy Populations | 13 |

| 8.2 | 2.1 I | Intention– to–treat population | 13 |
|--------|----------|------------------------------------------------|----|
| 8.2 | 2.2 | Safety population | 13 |
| 8.3 | Subg | group definitions | 13 |
| 8.4 | Trea | tment assignment and treatment groups | 13 |
| 9 Pat | ient D | Disposition | 13 |
| 10 De | mogra | aphics and Baseline characteristics | 14 |
| 11 Int | erim a | analysis and timing for analysis | 14 |
| 11.1 | Inter | im analysis | 14 |
| 11.2 | Time | points for analysis | 14 |
| 12 Fea | asibilit | ty and Efficacy Analysis | 15 |
| 12.1 | Meth | nod for analysis of endpoints | 15 |
| 12 | .1.1 | Analysis of feasibility endpoints | 15 |
| 12 | .1.2 | Analysis of efficacy endpoints | 15 |
| 12 | .1.3 | Analysis of subgroups | 15 |
| 12 | .1.4 | Covariate adjusted analysis | 15 |
| 12.2 | Assu | Imptions for analysis | 15 |
| 12.3 | Meth | nods for handling of missing data and outliers | 15 |
| 12.4 | Mult | iple comparisons | 16 |
| 12.5 | Mult | i–centre studies | 16 |
| 13 Saf | ety an | nalysis | 16 |
| 13.1 | Adve | erse events (AE) | 16 |
| 13.2 | Deat | ths or serious adverse events (SAE) | 16 |
| 14 Pre | esenta | tion of analysis | 17 |
| 15 PF | FEDEN | CFS | 23 |

### 4 GLOSSARY of Terms and Abbreviations

AE Adverse event
AF Atrial Fibrillation
BMI Body Mass Index
BP Blood Pressure

CHADS Score for estimating AF stroke risk

CI Confidence Interval
DBP Diastolic Blood Pressure

DC Direct Current

DCCV Direct Current Cardioversion

DSMC Data and Safety Monitoring Committee

ECG Electrocardiogram

FU Follow-up HR Heart Rate

IQR Interquartile Range

LA Left Atrial

LINQ Reveal LINQ cardiac monitoring system

LVEF Left Ventricular Ejection Fraction

Martal Health Composite Scale (SE 12)

MCS Mental Health Composite Scale (SF-12)

MI Myocardial infarction

BI Blinding Index OR Odds Ratio

PCI Percutaneous Coronary Intervention
PCS Physical Health Composite Scale (SF-12)
PROMS Patient Reported Outcome Measures

PVI Pulmonary Vein Isolation

QoL Quality of Life

R "R" Statistical Programming Software

SAE Serious Adverse Event SAP Statistical Analysis Plan

SF-12 Twelve item short form survey

SBP Systolic Blood Pressure SD Standard Deviation

#### 5 Introduction

This SAP has been written based on information from the study protocol version 2.0, dated 25/06/2019.

#### 5.1 Preface

Cardioversion with antiarrhythmic medication is commonly used as a first-line rhythm control strategy for patient with persistent atrial fibrillation (AF) despite having high recurrence and complication rates. Further options such as catheter ablation are considered once AF recurs. Patients with persistent AF undergoing catheter ablation are reported to have fewer symptoms and better quality of life than those undergoing DC cardioversion (DCCV) or optimal medical therapy. However, as yet this has not been subjected to a randomised, prospective, blinded clinical trial to measure the benefits of first-line AF ablation<sup>1</sup>.

### 5.2 Purpose of the analyses

The aim of a future main clinical trial would be to investigate whether patients undergoing DC cardioversion (DCCV) with the addition of a pulmonary vein isolation (PVI) cardiac ablation procedure with cryoablation for atrial fibrillation (AF) will have lower rates of AF recurrence than those treated by DCCV without a cardiac ablation procedure. The trial will also assess symptoms, quality of life, functional status and treatment satisfaction. This pilot study aims to validate the key study logistics with a view to optimising the methods to be used in a future main trial and will also give an initial assessment of efficacy outcomes.

## 6 Study objectives and design

## 6.1 Design

ORBITA-AF feasibility study is an internal pilot study. It is a randomised blinded controlled trial at two sites. Patients will be randomised to receive DCCV+PVI or DCCV alone. No information about the procedure will be transferred from catheterisation laboratory (cath lab) staff to recovery staff and cath lab staff will have no further contact with the patient during the study. Patients and other healthcare professionals will remain blinded to treatment allocation. If a future trial is determined to be feasible and no major changes to the design have been made from this pilot study, then pilot study patients will be included in the future main trial. This pilot study aims to recruit 20 patients.

## 6.2 Study objectives

The main hypotheses to be tested in a full trial of this nature would be that AF ablation reduces the recurrence of persistent AF and improves quality of life compared to acute treatment of heart rhythm by cardioversion and best medical therapy. Through this pilot study, the main objective is to assess operational aspects of the trial in order to optimise methods for a future main trial. In addition, descriptive analyses of study outcome measures will also be undertaken.

### 6.3 Feasibility Endpoints

- Protocol non-adherence (a) cross-over from one study group to the other, (b) do not receive randomised intervention.
- Recruitment rate (number recruited per month).
- Loss to follow-up at 12-months.
- Assessment of the success of the blinding procedure (i.e. blinding index).
- Data completeness.
- Key study logistics especially around the delivery of the intervention, including the use of a 'chaperone' to maintain blinding.
- Identifying barriers and facilitators to implementation.
- Assessment of the feasibility of the blinding SOP.
- Assessment of the acceptability of the interventions.
- Descriptive assessment of outcome measures for main trial (as below).

## **6.4 Efficacy Endpoints**

#### 6.4.1 Primary endpoint

• Recurrence of Persistent AF (AF episode lasting > 7 days) within 12 months.

#### 6.4.2 Secondary endpoints

- Death within 12 months.
- Hospital re-admission for any reason.
- Procedural-related complications.
- Bleeding events within 7 days of procedure.
- Requirement for repeat procedures within 12 months.
- Change in ejection fraction.
- Clinical success of procedure.
- Change in quality of life, as measured by SF-12 and AF-PROMS at 12 months.
- AF burden as measured on continuous monitoring.
- Antiarrhythmic drug use within 12 months.

## 6.4.3 Schedule of Assessment

| Assessment | Screening/ | Randomis | Treatment/ | Implant | Recovery | 6 weeks | 3 month | 12 month | Monthly | Registry |
|---|---|---|---|---|---|---|---|---|---|---|
| | pre- | ation | Procedure | | | (telephone) | | /EOS | downloads | |
| | admission | | | | | | (clinic) | (clinic) | | |
| Visit window | -14 days | Day 0 | Day 0 | Day 0 | | 42 days +/- 3 | +/- 7 days | +/- 2 weeks | | |
| | | | | | | days | | | | |
| Informed consent | Х | | | | | | | | | |
| Patient baseline characteristics | Х | | | | | | | | | |
| recorded: estimated AF | | | | | | | | | | |
| duration, LA dimensions (echo), | | | | | | | | | | |
| LVEF, Bloods, Medications, Age, | | | | | | | | | | |
| Sex, BP, CHADS VASC score, co- | | | | | | | | | | |
| morbidities, demographics, | | | | | | | | | | |
| weight, height, BMI. | | | | | | | | | | |
| Randomisation | | Х | | | | | | | | |
| DCCV only | | | Х | | | | | | | |
| DCCV plus Pulmonary Vein | | | Х | | | | | | | |
| Isolation | | | | | | | | | | |
| Telephone FU | | | | | | Х | | | | |
| Quality of life measures | Х | | | | | Х | Х | Х | | |
| Clinical FU | | | | | | Х | Х | Х | | |
| Loop recorder inserted | | | | Х | | | | | | |
| 12 lead ECG | | | | | Х | | Х | Х | | |
| Interrogation of loop recorder | | | | Х | | | Х | Х | Х | |
| Symptom questionnaires | Х | | | | | Х | Х | Х | | |
| Clinical status and mortality | | | | | | | | | | Х |
| data | | | | | | | | | | |

#### 6.4.4 Assessment of feasibility endpoints

Protocol non-adherence is defined as the proportion of patients in each randomised group who undergo the treatment that they were not randomised to as part of the index procedure, i.e. those randomised to DCCV only undergoing DCCV plus PVI, and those randomised to the DCCV plus PVI group who only undergo DCCV as part of the index trial procedure.

Recruitment rate will be defined as the total number of patients recruited divided by the number of months during which recruitment takes place.

Loss to follow-up will be defined as a) the number lost to follow-up at 12 months as a proportion of the number randomised. b) the number who do not consent to the collection of 5-year registry data as a proportion of the number randomised.

Data completeness will be defined as the number of subjects completing each assessment as a proportion of the total randomised. For this pilot study, analyses will be conducted on a complete case basis, and the level of missing data will be assessed to help inform as to best methods to use to handle potential missing data within a larger future trial.

Blinding index will be assessed as described by Bang et al (BI)<sup>2</sup>. Patients and staff will be asked to guess the treatment allocation and will answer DCCV, DCCV+PCI, or don't know. The BI is scaled to an interval of -1 to 1 with 1 being complete lack of blinding, 0 being perfect blinding and -1 indicating opposite guessing.

Other feasibility endpoints including assessing study logistics, identifying barriers and facilitators to implementation, and assessing the acceptability of the interventions will be assessed qualitatively, and hence will not be described further in the SAP.

#### 6.4.5 Assessment of primary and secondary efficacy endpoints

The primary endpoint is defined as the proportion of randomised patients with recurrent AF (AF episode lasting > 7 days) within 12 months, but outside of the initial 6-week blanking period (see section 8.1.2).

Secondary endpoints to be described are:

- Proportion dying within 12 months
- Proportion with hospital admission for any reason within 12 months
- Proportion with procedural-related complications defined as any AE that is deemed at least possibly related to intervention
- Proportion with bleeding events within 7 days of procedure
- Proportion with repeat procedures (any additional procedure for AF after the baseline index trial procedure(s)) within 12 months
- Change in ejection fraction from baseline at 12 months
- Proportion with clinical success of procedure
- Change in QoL at 12 months, as measured by SF-12 and AF-PROMS
- AF burden by 12 months
- Anti-arrhythmic drug use.

Clinical success will be defined as a 75% or greater reduction in the number of AF episodes as measured by the Reveal LINQ implant device within 12 months, but outside of the initial 6-week blanking period.

Change in QOL will be measured by the change in AF-PROMS summary scores and SF-12 PCS and MCS between screening and 12 months. SF-12 scores will be calculated as described in the appendix supplementary table 2<sup>3</sup>.

AF burden will be defined as the proportion of time in AF over the 12 months but outside of the initial 6-week blanking period, as measured by the Reveal LINQ implant device.

## 6.5 Level of significance

No hypothesis testing will be done for this pilot study.

For efficacy outcome measures we will use 80% one-sided confidence intervals to give an indication of whether the endpoint is likely to be of interest, an approach described by Cocks et al. for pilot trials<sup>4</sup>.

### 6.6 Sample size

The sample size of 20 subjects has been chosen as an achievable recruitment target that would enable assessment of feasibility of the study, and to confirm whether a larger trial could be conducted. At around 10% of a sample size required for a future main trial, this will also allow an initial assessment of the effectiveness of the intervention using a confidence interval approach<sup>4</sup>.

## 7 General Analysis Definitions

## 7.1 Study period and visit definitions

#### 7.1.1 Visits

Patients will be identified as suitable for the study by their usual clinical care provider. Patients referred for DC cardioversion or management of persistent AF will be screened for inclusion into the trial. Patients will give informed consent in pre-admission. Baseline characteristics, quality of life and symptom measures will be assessed at this point.

On the day of the procedure patients will be randomised to DCCV or Pulmonary Vein Isolation plus DCCV. LINQ will be inserted during the procedure. Patients will be followed up at 6 weeks by telephone for quality of life and symptom measures.

Patients will return to the clinic at 3 months (clinical follow-up, 12 lead ECG, repeat QOL and symptom measures) and at 12 months (clinical follow-up, 12 lead ECG and symptoms). Monthly remote interrogation of the loop recorder will measure burden of AF (time in AF) and duration of episodes.

Patients who consent will remain within an observational registry for 5 years following the end of the trial. This long-term passive follow-up will track patient mortality and clinical status from

routinely collected clinical data. No intervention or investigations will be performed as part of this long term follow up.

Data from this pilot study will be analysed at 12 months to allow assessment of feasibility for a larger trial, and patients who complete the 12-month follow-up visit and consent will continue in registry follow-up for 5 years post procedure.

#### 7.1.2 Study Scheme Diagram



### 7.2 Study Populations

#### 7.2.1 Intention- to-treat population.

Results will be presented on an intention to treat basis with all randomised patients analysed according to the group they were assigned to, regardless of whether the treatment was received or whether the protocol was adhered to.

#### 7.2.2 Safety population

The safety population will consist of all randomised patients who received the allocated treatment.

### 7.3 Subgroup definitions

No subgroup analysis will be undertaken.

### 7.4 Treatment assignment and treatment groups

Patients will be randomised on a 1:1 basis to either DCCV alone or DCCV + PVI. Block randomisation is used with randomly varying block sizes of length 2, 4, and 6. Randomisation will not be stratified by any factors. The allocation algorithm is written by the study statistician using R (randomizeR package). Details of the randomisation method and validation details are stored in a separate document which can be accessed by the trial statistician and the database manager.

The randomisation list will then be uploaded to the study database (REDCap). When a patient has been screened and has met all of the entry criteria in order to be eligible for trial participation, the unblinded investigator will go to the randomisation module on the database and complete the randomisation form. Once complete, the allocation (which is next in the sequence on the randomisation list) will be revealed to the unblinded investigator.

## 8 Patient Disposition

Participants will be those referred for either cardioversion for persistent AF (> 7 days) or catheter ablation of persistent AF. Inclusion/exclusion criteria are detailed in the protocol (section 7). Numbers of patients screened, excluded prior to randomisation by reason and overall, randomised and completing each phase of the study will be shown by treatment groups and overall following the Consort structure.

## 9 Demographics and Baseline characteristics

Demographic and baseline (screening data) will be:

- 1. Age
- 2. Sex
- 3. Ethnicity
- 4. BMI
- 5. SBP
- 6. DBP
- 7. HR
- 8. AF duration
- LVEF
- 10. Diabetes
- 11. Current Smoking
- 12. Hypertension
- 13. Hypercholesterolaemia
- 14. Previous MI
- 15. Previous PCI

Demographic and baseline data will be summarised by randomisation group and overall. For continuous data the number of subjects, mean, SD, median and interquartile range will be shown. For categorical data number and percentage will be shown. No formal testing will be performed for the comparison of baseline characteristics.

## 10 Interim analysis and timing for analysis.

## 10.1 Interim analysis

On completion of the 6-week blinding period of the last patient to be enrolled into the pilot study, an interim analysis will be performed, including endpoints assessed from baseline to 6-weeks. No other interim analyses are panned prior to the completion of the study, unless specifically requested by the DSMC.

The main analysis will take place at the end of this pilot study and this information will be used to inform decisions regarding procedure to a main future trial. Patients will be followed up for 12 months regardless of interim analysis results.

## 10.2 Time points for analysis.

The DSMC will monitor patient safety and will meet prior to initiation of the study, after the recruitment of 4 patients and then at 3 monthly intervals. All other analysis described in this SAP will take place at the end of this pilot study.

## 11 Feasibility and Efficacy Analysis

## 11.1 Method for analysis of endpoints

#### 11.1.1 Analysis of feasibility endpoints

Proportions will be shown along with the number with each binary endpoint and total number.

The recruitment rate will be shown overall as the total number of patients recruited divided by the number of months.

Data completeness will be assessed as the numbers with and without data recorded and the proportion with complete data for each treatment group and overall.

For the blinding index, the number and percentage with each response will be given for each treatment arm. The blinding index will be reported for each group.

Other feasibility endpoints, including assessment of key study logistics, and the feasibility of blinding SOP, acceptability of interventions, will be assessed more qualitatively, and hence will not be described further in this SAP.

#### 11.1.2 Analysis of efficacy endpoints

Categorical variables will be shown as the number with each endpoint and total number in each group along with the proportion. Odds ratios and 80% one-sided exact confidence intervals will also be shown as an assessment of efficacy, an approach described by Cocks et al<sup>4</sup>.

For continuous variables mean, SD, and number of patients with available data will be presented along with estimated mean difference between trial arms and 80% one-sided confidence intervals.

For AF burden (proportion of time in AF), median and IQR will also be reported.

#### 11.1.3 Analysis of subgroups

There is no plan to conduct any subgroup analyses.

#### 11.1.4 Covariate adjusted analysis

No covariate adjustment will take place.

### 11.2 Assumptions for analysis.

For continuous efficacy outcomes, confidence intervals for differences will be constructed assuming a normal distribution. Normality of distribution for continuous variables is hard to assess with such a small number of subjects in this pilot trial and so will not have much value.

## 11.3 Methods for handling of missing data and outliers

This pilot study will assess data completeness to inform decisions about missing data for a future main trial. Analysis will use all patients with available endpoint data. The level of missing data will be tabulated for each outcome, presenting the number of subjects with a data record and number with missing data, separately by trial arm.

### 11.4 Multiple comparisons

No adjustment for multiple comparisons will be made.

#### 11.5 Multi-centre studies

No adjustment will be made for centre in this pilot study.

## 12 Safety analysis

## 12.1 Adverse events (AE)

AEs will be summarised using counts and percentages. The number of subjects having at least one AE will be presented overall and tabulated by treatment. The number of subjects with AEs of mild/moderate/severe intensity will be shown overall and by treatment using the maximum severity experienced for each patient. The total number of AEs for each treatment, allowing multiple events per patient, will also be presented.

#### 12.2 Deaths or serious adverse events (SAE)

SAEs will be listed separately along with details of the treatment and whether the event is unexpected and whether it is thought to be related to the treatment.

## 13 Presentation of analysis

Results will be presented as follows.

Figure 1: Consort flow diagram



Table 1: Tables of demographic and baseline characteristics, overall and by treatment group

| | | Treatme | nt group | |
|---|---|---|---|---|
| | | DCCV<br>(N=) | DCCV +PVI<br>(N=) | Combined<br>(N=) |
| Age (years) | | Mean (SD) | Mean (SD) | Mean (SD) |
| Sex | Female | n/N (%) | n/N (%) | n/N (%) |
| sex | Male | n/N (%) | n/N (%) | n/N (%) |
| | Asian | n/N (%) | n/N (%) | n/N (%) |
| | Black | n/N (%) | n/N (%) | n/N (%) |
| Ethnicity | Mixed | n/N (%) | n/N (%) | n/N (%) |
| | Other | n/N (%) | n/N (%) | n/N (%) |
| | White | n/N (%) | n/N (%) | n/N (%) |
| BMI (kg/m²) | | Mean (SD) | Mean (SD) | Mean (SD) |
| SBP (mmHg | g) | Mean (SD) | Mean (SD) | Mean (SD) |
| DBP (mmH | g) | Mean (SD) | Mean (SD) | Mean (SD) |
| HR (bpm) | | Mean (SD) | Mean (SD) | Mean (SD) |
| AF duratio | n (months) | Median [IQR] | Median [IQR] | Median [IQR] |
| | | Mean (SD) | Mean (SD) | Mean (SD) |
| Left Ventri<br>(%) | cular Ejection Fraction | Median [IQR] | Median [IQR] | Median [IQR] |
| | T | Mean (SD) | Mean (SD) | Mean (SD) |
| Current | Non- smoker | n/N (%) | n/N (%) | n/N (%) |
| Smoking | Previous smoker Current smoker | n/N (%) | n/N (%) | n/N (%) |
| Diabetes | Current smoker | n/N (%)<br>n/N (%) | n/N (%)<br>n/N (%) | n/N (%)<br>n/N (%) |
| Renal insuf | ficiency | n/N (%) | n/N (%) | n/N (%) |
| | vascular disease | n/N (%) | n/N (%) | n/N (%) |
| Hypertensi | on | n/N (%) | n/N (%) | n/N (%) |
| Hyperchole | esterolaemia | n/N (%) | n/N (%) | n/N (%) |
| Previous st | roke | n/N (%) | n/N (%) | n/N (%) |
| Previous M | II | n/N (%) | n/N (%) | n/N (%) |
| Previous Po | CI | n/N (%) | n/N (%) | n/N (%) |

Table 2: Feasibility endpoints

| | Treatme | | |
|--------------------------------|-----------|-----------|----------|
| | DCCV | DCCV +PVI | Combined |
| | (N=) | (N=) | |
| Proportion crossing over | | | - |
| | n/N (%) | n/N (%) | |
| Proportion with off-protocol | n/N (%) | n/N (%) | n/N (%) |
| deviation | | | |
| Recruitment rate | | | Rate |
| (patients per month) | - | - | |
| Loss to follow-up at 12 months | n/N (%) | n/N (%) | n/N (%) |
| Not consenting to 5-year | n/N (%) | n/N (%) | n/N (%) |
| registry data follow-up | , (*-1 | , ( | , (-, |
| Blinding index | | | |
| Staff - post procedure | | | |
| DCCV | n11 (p11) | n21 (p21) | - |
| DCCV + PCI | n12 (p12) | n22 (p22) | - |
| Don't know | n13 (p13) | n23 (p23) | - |
| Total | N1 | N2 | - |
| Blinding index | ВІ | BI | - |
| Patients - post procedure | | | |
| DCCV | n11 (p11) | n21 (p21) | - |
| DCCV + PCI | n12 (p12) | n22 (p22) | - |
| Don't know | n13 (p13) | n23 (p23) | - |
| Total | N1 | N2 | - |
| Blinding index | ВІ | BI | - |
| Patients - 6 weeks | | | |
| DCCV | n11 (p11) | n21 (p21) | - |
| DCCV + PCI | n12 (p12) | n22 (p22) | - |
| Don't know | n13 (p13) | n23 (p23) | - |
| Total | N1 | N2 | - |
| Blinding index | BI | BI | - |
| Patients - 3 months | | | |
| DCCV | n11 (p11) | n21 (p21) | - |
| DCCV + PCI | n12 (p12) | n22 (p22) | - |
| Don't know | n13 (p13) | n23 (p23) | - |
| Total | N1 | N2 | - |
| Blinding index | BI | BI | - |

**Table 3: Data completeness** 

| | Treatme | nt group | |
|---|---|---|---|
| | DCCV<br>(N=) | DCCV +PVI<br>(N=) | Total |
| Primary Endpoint data | N1 | N1 | N1 |
| (Persistent AF) | N2 | N2 | N2 |
| | % with data | % with data | % with data |
| SF12 | | | |
| 3 months | N1 | N1 | N1 |
| | N2 | N2 | N2 |
| | % with data | % with data | % with data |
| 12 months | N1 | N1 | N1 |
| | N2 | N2 | N2 |
| | % missing | % missing | % with data |
| AF-PROMS | | | |
| 3 months | N1 | N1 | N1 |
| | N2 | N2 | N2 |
| | % with data | % with data | % with data |
| 12 months | N1 | N1 | N1 |
| | N2 | N2 | N2 |
| | % with data | % with data | % with data |
| Loop recorder interrogation performed | | | |
| 3 months | | | |
| | N1 | N1 | N1 |
| | N2 | N2 | N2 |
| 12 Months | % with data | % with data | % with data |
| | N1 | N1 | N1 |
| | N2 | N2 | N2 |
| | % with data | % with data | % with data |
| Patients completing all | N1 | N1 | N1 |
| study assessments | N2 | N2 | N2 |
| | % with data | % with data | % with data |

N1= Number with data recorded

N2=Number with missing data

Table 4: Primary and Secondary Efficacy Endpoint analysis (ITT population)

| | Treatme | | |
|---|---|---|---|
| | Placebo | Active | OR (80% CI) |
| | N= | N= | |
| Recurrent AF within 12 months | n/N (%) | n/N (%) | |
| Death within 12 months | n/N (%) | n/N (%) | |
| Hospital admission within 12 months | n/N (%) | n/N (%) | |
| Procedural-related complications | n/N (%) | n/N (%) | |
| Bleeding events within 7 days | n/N (%) | n/N (%) | |
| Requirement for repeat procedures within 12 months | n/N (%) | n/N (%) | |
| Clinical success of procedure | n/N (%) | n/N (%) | |
| AF drug use within 12 months | n/N (%) | n/N (%) | |
| | Placebo<br>N= | Active<br>N= | b (80% CI) |
| Change in ejection fraction at 12 months | Mean (SD) | Mean (SD) | |
| AF-Burden | Median [IQR]<br>N | Median [IQR]<br>N | |
| | Mean (SD) | Mean (SD) | |
| Change in QoL score at 12 months: SF-12 MCS | Mean (SD)<br>N | Mean (SD) | |
| SF-12 PCS | Mean (SD)<br>N | Mean (SD)<br>N | |
| AF-PROMS | Mean (SD)<br>N | Mean (SD)<br>N | |

Table 5: Safety analysis – adverse events (safety population)

| | | Treatment group | |
|---|---|---|---|
| | | Placebo<br>N= | Active<br>N= |
| Number of patients experiencing an AE within a year | | n/N (%) | n/N (%) |
| Maximum severity AE experienced | Mild | n/N (%) | n/N (%) |
| | Moderate | n/N (%) | n/N (%) |
| | Severe | n/N (%) | n/N (%) |
| Total number of AEs across patients | | n | n |

Table 6: SAE listing

| SAE<br>number | Patient<br>ID | SAE term<br>(MedDRA) | SAE<br>severity | Expected/<br>unexpected | Treatment group | Details of treatment | Related to treatment? |
|---|---|---|---|---|---|---|---|
| 1 | | | | | | | |
| 2 | | | | | | | |
| 3 | | | | | | | |
| 4 | | | | | | | |
| ••• | | | | | | | |

#### 14 REFERENCES

- 1) January, C. T., Wann, L. S., Alpert, J. S., Calkins, H., Cigarroa, J. E., Cleveland, J. C., Jr.American College of Cardiology/American Heart Association Task Force on Practice, G. (2014). 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. *J Am Coll Cardiol, 64*(21), e1-76.
- 2) Bang H, Ni L, Davis CE (2004). Assessment of blinding in clinical trials. Controlled Clinical Trials, 25(2): 143-156.
- 3) Gonzalez-Chica DA, Dal Grande E, Bowden J, Musker M, Hay P, Stocks N (2017). Are we reducing the risk of cardiovascular disease and improving the quality of life through preventive health care? Results of a population-based study in South Australia. Preventive medicine, 99,164-170.
- 4) Cocks K, Togerson DJ (2013), Sample size calculations for pilot randomized trials: a confidence interval approach. Journal of Clinical Epidemiology, 66:197-201.